CLINICAL TRIAL: NCT02936115
Title: A Multicenter, Randomized, Single-Blind Study Comparing the Clinical Outcomes of TruSkin® and an Active Comparator for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: TruSkin®: Study for the Treatment of Chronic Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Osiris decision
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Osiris Protocol 351
Record Dates: First submitted 2016-09-20; First posted 2016-10-18 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TruSkin® (Experimental): Cryopreserved skin allograft
  Interventions: Other: TruSkin®
- Wound Cover (Active Comparator): Active Comparator for Diabetic Foot Ulcers
  Interventions: Other: Wound Cover

INTERVENTIONS:
Other: TruSkin®
  Arms: TruSkin®
Other: Wound Cover
  Arms: Wound Cover

SUMMARY:
The purpose of this study is to compare the clinical outcomes of TruSkin® and an Active Comparator in patients with chronic diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years and 80 years of age inclusive, as of the date of screening
2. Confirmed diagnosis of Type 1 or Type 2 Diabetes
3. An Index Ulcer that is chronic (defined as present for > 4 weeks, but not present for more than 52 weeks at the Screening Visit)
4. Index Ulcer is located below the malleolus
5. The Index Ulcer is a Diabetic Foot Ulcer (DFU) greater than 3 cm2, inclusive, at the Screening Visit
6. The longest length and longest width measurements for the Index Ulcer are no less than 1 cm each at the Screening Visit
7. The Index Ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone, or joint capsule
8. Wound is free of necrotic debris
9. Patient has adequate circulation to the foot as documented by ABI or TBI

Exclusion Criteria:

1. Index Ulcer is of non-diabetic pathophysiology
2. Gangrene is present on any part of the affected foot
3. Index Ulcer is over a Charcot deformity
4. Patient is currently receiving dialysis or planning to go on dialysis
5. Patient has a glycated hemoglobin A1c (HbA1c) level of >12%
6. Chronic oral steroid use >7.5 mg daily for longer than 3 months at the time of screening
7. Patient is receiving IV corticosteroids, immunosuppressive or cytotoxic agents at the time of screening
8. Requiring intravenous (IV) antibiotics to treat the index wound infection at the time of screening
9. Patient has an ulcer within 5 cm of the Index Ulcer identified for study consideration
10. Patient is Human Immunodeficiency Virus (HIV) positive or has Acquired Immune Deficiency Syndrome (AIDS)
11. Current evidence of cellulitis, or other evidence of infection including fever or pus drainage from the wound site
12. Current evidence of osteomyelitis or history of osteomyelitis within 30 days of screening
13. Patient has active malignancy other than non-melanoma skin cancer
14. Patient's Index Ulcer has decreased by ≥ 20% during 1-week screening period
15. Patient's random blood sugar is > 450 mg/dl at screening
16. Patient is unable to properly off-load the index wound as a part of standard of care
17. Patient has untreated alcohol or substance abuse at the time of screening
18. Pregnant women and women who are breastfeeding
19. Patient is currently enrolled or participated in another investigational device, drug, or biological trial within 30 days of screening
20. Patient has had within the last 30 days, or is currently undergoing, or is planning for wound treatments with growth factors, living skin, dermal substitutes or other advanced biological therapies
21. Patient is an employee, or an immediate family member of an employee, of the sponsor company or site research staff conducting the study
22. Patients who have already been randomized in Protocol 351 at any center may not be considered for screening or for re-entry into the trial at any center, even after the End of Study Visit
23. Patients with a history of poor compliance, or an unwillingness or inability to adhere to the requirements of the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients that achieve a 50% or greater reduction in wound size by 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Proportion of patients that achieve complete closure of the index wound by 12 weeks | 12 weeks
Proportion of Patients that achieve a 50% or greater reduction in wound size by 4 weeks | 4 weeks
Time to initial wound closure | Up to 84 days
Number of product applications | Up to 84 days
Number of AEs | Up to 84 days
Number of patients with worsening of index wound defined by ≥ 50% increase in wound size | Up to 84 days

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Florida City, Florida
  - Illinois City, Illinois
  - Michigan, Michigan
  - Texas City, Texas
  - Virginia City, Virginia

IPD SHARING:
Plan to Share IPD: No